CLINICAL TRIAL: NCT03709342
Title: A Pharmacodynamic and Pharmacokinetic Study of CM4620 Injectable Emulsion (CM4620-IE) in Patients With Acute Pancreatitis
Brief Title: A PK/PD Study of CM4620-IE in Patients With Acute Pancreatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CalciMedica, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM4620-202
Record Dates: First submitted 2018-10-11; First posted 2018-10-17 (Actual); Results first posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-02

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Patients (Experimental)
  Interventions: Drug: CM4620-IE

INTERVENTIONS:
Drug: CM4620-IE — single IV infusion on Day 1 over 4 hours

SUMMARY:
This open-label study will evaluate the pharmacodynamic and pharmacokinetic profile of CM4620-IE in patients with acute pancreatitis. The first five (5) patients will receive ≤ 2.08 mg/kg of CM4620-IE by continuous IV infusion on Day 1. If necessary, up to an additional 4 patients may be treated at a different dose of CM4620-IE as determined by the obtained PK and PD data. The infusion of CM4620-IE will start within 12 hours from the time the patient or LAR provides informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of acute pancreatitis established by the presence of abdominal pain consistent with acute pancreatitis, and 1 of the following 2 criteria:

   1. Serum lipase and/or serum amylase > 3 times the upper limit of normal (ULN);
   2. Characteristic findings of acute pancreatitis on abdominal imaging;
2. Adults ≥ 18 years of age;
3. A female patient of child-bearing potential who is sexually active with a male partner must be willing to practice acceptable methods of birth control for 365 days after the last dose of CM4620-IE;
4. A male patient who is sexually active with a female partner of childbearing potential must be willing to practice acceptable methods of birth control for 365 days after the last dose of CM4620-IE and must not donate sperm for 365 days;
5. Willing and able to, or have a legal authorized representative (LAR) who is willing and able to, provide informed consent to participate, and cooperate with all aspects of the protocol.

Exclusion Criteria:

1. Any concurrent clinical condition that a study physician believes could potentially pose an unacceptable health risk to the patient while involved in the study or may limit expected survival to < 6 months;
2. Suspected presence of cholangitis in the judgment of the treating investigator;
3. Any malignancy being treated with chemotherapy or immunotherapy;
4. Any autoimmune disease being treated with immunosuppressive medication or immunotherapy (Section 5.3 for list of prohibited medications);
5. History of:

   1. Chronic pancreatitis, pancreatic necrosectomy, or pancreatic enzyme replacement therapy;
   2. Biopsy proven cirrhosis, portal hypertension, hepatic failure/hepatic encephalopathy;
   3. Known hepatitis B or C, or HIV;
   4. History of organ or hematologic transplant;
   5. Myocardial infarction, revascularization, cardiovascular accident (CVA) in the 30 days prior to Day 1;
6. Current renal replacement therapy;
7. Current known abuse of cocaine or methamphetamine;
8. Known to be pregnant or are nursing;
9. Participated in another study of an investigational drug or therapeutic medical device in the 30 days prior to Day 1;
10. History of allergy to eggs or known hypersensitivity to any components of CM4620-IE;
11. Prior treatment with CM4620-IE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-01-06 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2019-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudarshan Hebbar, MD, Study Director — CalciMedica, Inc.
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Patients
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Exploratory: Percentage Change in IL-2 Production Relative to Pre-dose Values
Description: Outcome assessed the percent change in IL-2 production after the administration of a single dose of CM4620-IE as compared to baseline production, for all patients enrolled. This measurement was to explore if there was a change in IL-2 levels with acute pancreatitis after the administration of a single dose of CM4620-IE.
Time Frame: Predose to 30 minutes post dose
Population: The final analysis set consisted of pre-dose to Discharge samples for 4 patients, due to logistical issues in timely assaying of the samples.
Measure: Mean (Standard Error); unit: percentage of change in IL-2 production
Arm/Group | All Patients
Number analyzed (Participants) | 4
percentage of change in IL-2 production | -55.5 (5.8)

2. Secondary Outcome: The Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]
Description: The number of participants who experienced treatment-emergent adverse events (TEAEs) with Investigator-specified relationship to CM4620-IE and assessment of severity.
Time Frame: From baseline through 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 7
Participants | 3

3. Secondary Outcome: Pharmacokinetics (CMax of CM4620): Day 1, 30 Minutes Post End-of-infusion
Time Frame: Days 1, 2, 5, 10 and 30 or at discharge if earlier than day 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms/mL
Arm/Group | All Patients
Number analyzed (Participants) | 7
Nanograms/mL | 791 (47)

4. Secondary Outcome: Pharmacokinetics (Plasma Concentration of CM4620): Day 2, 20-hr Post End-of-infusion
Description: Time points for sampling of plasma for bioanalysis of CM4620, blood for PD analysis (stimulated IL-2 release), and serum for cytokine analysis were chosen to capture the expected maximal plasma concentration (Cmax) on Day 1 and times close to the minimum plasma concentration (Cmin) on subsequent days.
Time Frame: Day 2
Population: Samples were only received for analysis for 5 patients for day 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ng/mL
Arm/Group | All Patients
Number analyzed (Participants) | 5
Ng/mL | 109 (49)

5. Secondary Outcome: Pharmacokinetics (Plasma Concentration of CM4620): Day 10 or Discharge
Time Frame: Day 10, or day of discharge
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ng/mL
Arm/Group | All Patients
Number analyzed (Participants) | 7
Ng/mL | 76 (46)

6. Secondary Outcome: Pharmacokinetics (Plasma Concentration of CM4620): Day 30
Time Frame: Day 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ng/mL
Arm/Group | All Patients
Number analyzed (Participants) | 7
Ng/mL | 56 (32)

7. Secondary Outcome: Baseline Levels of IL-6
Description: Included plasma samples collected 1 hour prior to the study drug administration
Time Frame: Baseline
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | All Patients
Number analyzed (Participants) | 7
pg/mL | 46.04 (26.3)

8. Secondary Outcome: Day 1: 30 Minutes Post-infusion IL-6 Levels
Time Frame: Day 1
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | All Patients
Number analyzed (Participants) | 7
pg/mL | 40.83 (23.29)

9. Secondary Outcome: Day 2: 20-hr Post Infusion IL-6 Levels
Time Frame: Day 2
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | All Patients
Number analyzed (Participants) | 6
pg/mL | 24.8 (12.4)

10. Secondary Outcome: Post-infusion IL-6 Levels at Discharge
Description: This sample was drawn immediately prior to discharge from hospitalization, and ranged from day 2 through day 9.
Time Frame: Assessed at Discharge, between 2 and 9 days.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | All Patients
Number analyzed (Participants) | 7
pg/mL | 13.9 (2.0)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 90 days per subject, from the start of dosing until the 30-day follow-up.
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 3/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=7)
Acute Pancreatitis (Gastrointestinal disorders) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=7)
Melaena (Gastrointestinal disorders) | 1 (1)
Bursitis (Skin and subcutaneous tissue disorders) | 1 (1)
Acute Pancreatitis (Gastrointestinal disorders) | 1 (1) — This event is also captured as an SAE
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alcohol Withdrawal Syndrome (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) — This event is also captured as an SAE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/42/NCT03709342/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/42/NCT03709342/SAP_001.pdf